CLINICAL TRIAL: NCT07127588
Title: Continuing Education of General Practitioners in Clinical Ultrasound - Ultrasound Simulation or Traditional Ultrasound Training?
Brief Title: Ultrasound Simulation or Traditional Ultrasound Training for General Practitioners?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Nordsim (Unknown)
Responsible Party: Principal Investigator, Julie Jepsen Strøm, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 262-1
Record Dates: First submitted 2025-07-27; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Ultrasound Training
Keywords: Point-of-care ultrasound; Clinical ultrasound; Education; General practitioners; Simulation; Randomised controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation (Experimental): General practitioners allocated to the intervention arm will participate in the POCUS course with hands-on training on an ultrasound simulator which can portrait both the normal reference and pathology at hands-on teaching seminars.
  Interventions: Other: Simulation based clinical ultrasound education
- Healthy volunteers (Active Comparator): General practitioners allocated to the control arm will participate in the POCUS course with hands-on training on healthy volunteers and pathology presented as still pictures and videos at hands-on teaching seminars.
  Interventions: Other: Traditional ultrasound education

INTERVENTIONS:
Other: Simulation based clinical ultrasound education — At the two hands-on teaching seminars, GPs in the intervention arm will receive training in five different clinical ultrasound examinations using an ultrasound phantom and an ultrasound simulator (Simbionix U/S Mentor). At the start of the first course day (8 hours), three basic modules will be conducted on the simulator, aimed at training hand-eye coordination and developing fundamental skills in probe movement, enhancing three-dimensional perception, and learning to use the various settings on the ultrasound simulator to achieve optimal imaging. At the first course day, the five clinical ultrasound examinations will be trained through a total of 13 simulation cases. On the second course day (4 hours), the participants will repeat the 13 simulation cases.
  Arms: Simulation
Other: Traditional ultrasound education — At the two hands-on teaching seminars, GPs in the control arm will receive training in five different clinical ultrasound examinations as according to an established and validated training program. At the start of the first course day (8 hours), the five clinical ultrasound examinations will be trained using healthy volunteers and still pictures for visualizing pathology. On the second course day (4 hours), the participants will train by repeating the five clinical ultrasound examinations on healthy volunteers.
  Arms: Healthy volunteers

SUMMARY:
The goal of this study is to compare two different educational methods for training general practitioners (GPs) in point-of-care ultrasound. The main question it aims to answer is:

- Does the use of ultrasound phantoms and simulators result in superior post-course ultrasound skills compared to traditional training methods involving healthy volunteers? Researchers will compare a group trained with traditional methods (scanning healthy volunteers) to a group trained using ultrasound phantoms and simulators to see if the different training methods result in different levels of ultrasound proficiency.

Participants will:

* Be 24 general practitioners randomized into two groups of 12.
* Receive training in five clinical ultrasound examinations: 1) Aortic abdominal aneurism, 2) gallstones, 3) pleural effusion, 4) hydronephrosis, and 5) free fluid in the abdomen (FAST scan).
* Begin with e-learning, followed by two in-person teaching seminars.
* Train at their clinics between course days: first on healthy volunteers, then on indicated patients.
* Upload scans to an online learning platform and receive feedback from instructors.
* Be assessed after 90 days using the validated Objective Structured Assessment of Ultrasound Skills (OSAUS) tool, with blinded evaluators.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be a postgraduate medical doctor specialized in general medicine/family medicine (general practitioner).
* The participant must have access to an ultrasound device during the study period.

Exclusion Criteria:

* General practitioners who have already participated in a basic point-of-care ultrasound education for general practitioners.
* General practitioners with potential conflicts of interest.
* Individuals with no signed informed consent to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
Mean OSAUS sum score across all five POCUS applications (min-max: 7-35) | At the third teaching seminar (day 90)
  Scanning competence is assessed similarly in the two groups by ultrasound expert reviewers blinded to participant allocation. The reviewers will use the OSAUS score, which consists of 7 items. Each item is rated using a Likert Scale with five points (1-5) giving a minimum score of 7 and maximum of 35 for each POCUS application.

CONTACTS AND LOCATIONS:
Locations (1):
- NordSim, Aalborg, Denmark